CLINICAL TRIAL: NCT00798733
Title: A Multicenter Prospective Cohort Study of Sacral Fractures Using Patient Based and Objective Outcomes
Brief Title: Study of Sacral Fractures Using Patient Based and Objective Outcomes
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Foundation of Orthopedic Trauma (Other)
Responsible Party: Sponsor
Other Study IDs: H-27355
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Sacrum Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-Operative: Surgeon treated the patient non-operatively
- Operative: Surgeon treated the patient operatively

SUMMARY:
The purpose of this study is to define the outcomes, both patient based and radiographic, for sacral fractures based upon injury pattern, displacement, and treatment. This will aid the orthopaedist in determining the best course for those patients with mild to moderate displacement. Multiple centers will be included and not asked to change their protocols for management. The prospective evaluation will gather specific data points on mechanism of injury, displacements, position at union, and disease specific and general health outcomes.

DETAILED DESCRIPTION:
There is wide variation in the current treatment of pelvic ring trauma. This divergence in practice patterns includes the use of either operative or non-operative care for the same fractures. Sacral fractures are the most commonly observed posterior pelvic ring injury and comprise up to 75% of cases reported at most institutions. The optimal and appropriate treatment of these fractures is vigorously debated despite the common goal of improving patient outcomes. While significant posterior pelvic displacement is universally considered an appropriate operative indication in healthy individuals, the threshold for "significant" is poorly defined and difficulty to accurately measure. Further, lesser and minimal displacement patterns are currently being treated operatively and non-operatively, depending on the institution and the experience of the surgeon, and without adequate guidelines. This lack of consensus in the treatment of sacral fractures is due to a poor understanding of patient outcomes following operative and non-operative treatment, a poor understanding of how the morbidities associated with a specific treatment affect patient outcome, and a lack of data that allows any meaningful comparison of operative and non-operative treatment.

The purpose of this study is to define the patient-based and radiographic outcomes of sacral fractures based on injury pattern, fracture displacement, and treatment method. We anticipate that minimally displaced fractures will be treated non-operatively and significantly displaced fractures will be treated operatively by most centers. There will also be a group of patients with displacements that are treated operatively or non-operatively by different surgeons. We will document the outcomes for all three groups, and compare the outcomes of operative and nonoperative management for the middle (overlap) group. This will aid the orthopaedist in determining the best treatment courser for those patients based on displacement. Fourteen centers have agreed to participate with four already actively recruiting. The prospective evaluation will gather specific data points on mechanism of injury, displacements, position at union, and disease specific and general health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old and <=80 years old
* Unilateral sacral fractures
* Informed consent obtained
* Patient is English speaking

Exclusion Criteria:

* APC injuries
* Zone 3 sacral fractures
* Unable to comply with outcome measures, postoperative rehabilitation protocols or instructions (e.g. head injured or mentally impaired)
* Unlikely to follow-up in surgeon's estimation
* Incarcerated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through the Emergency Department or Orthopaedic Clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2017-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Majeed Pelvic Score | Obtained preoperatively and at 3, 6, 9, 12, and 24 month follow-ups
SMFA | Obtained preoperatively and at 3, 6, 9, 12, and 24 month follow-ups
VAS | Obtained preoperatively and 24 hours, 1, 3, and 6 weeks 3, 6, 9, 12, and 24 month follow-ups

SECONDARY OUTCOMES:
Radiographic displacement | Union

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta, MD, Principal Investigator — Boston University
Locations (14):
- United States (13):
  - Indiana University, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Missouri-Univerisity hospital, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma/ Health Science, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Orthopaedic Specialty Associates Fort Worth, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
- QEII Health Science Center-NHI, Halifax, Canada